CLINICAL TRIAL: NCT00832845
Title: Cognitive Behavioral Social Skills Training for Patients With Late-Life Schizophrenia: a Pilot Study
Acronym: CBSST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Tarek Rajji, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 066/2008
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
Keywords: Late-life schizophrenia (LLS); Cognitive Behavioural Social Skills Training (CBSST); Randomized
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBSST plus treatment as usual (Experimental): Subject randomized to the CBSST Group arm will attend 2 hour weekly Cognitive Behavioural Social Skills therapy sessions for 9 months. They will also be attending follow-up assessments q 4 months.
  Interventions: Behavioral: CBSST plus treatment as usual
- Treatment as Usual Group (Active Comparator): Subjects randomized to the Treatment as Usual Group Arm will continue with their regular psychiatric treatment for 1 year. Like the CBSST Group Arm, they will have follow up assessments q 4 months. After completing the Treatment as Usual Group arm, they will automatically continue on with the CBSST Group Arm.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: CBSST plus treatment as usual — Patients will receive CBSST in addition to their regular treatment for 36 weeks.
  Arms: CBSST plus treatment as usual
Behavioral: Treatment as usual (TAU) — Patients will receive their regular treatment for 36 weeks without CBSST. TAU consists of the standard care that patients receive, including routine visits and contacts with their physicians and clinicians.
  Arms: Treatment as Usual Group

SUMMARY:
Schizophrenia is associated with significant cognitive and functional deficits. As patients with schizophrenia grow older, the impact of these deficits at a personal and public health level is likely to increase. Cognitive Behavioral and Social Skills Training (CBSST) is a recently developed group therapy that increased the frequency of social activities among middle-aged patients with schizophrenia. It also increased cognitive insight, a measure of the ability to reduce confidence in aberrant beliefs. To date, CBSST has not been studied in late-life schizophrenia. In addition, its impact on medications management, an instrumental function that is particularly salient in late life, and its interactions with cognition are largely unknown. Thus, we propose to study the efficacy of CBSST in improving social skills and medications management in patients with late-life schizophrenia, and to study the interactions between the patients' cognitive characteristics and their response to CBSST.

Previous studies show that cognitive deficits are strong predictors of response to CBSST. Cognitive Remediation Treatments (CRTs) have been shown to improve cognition in patients with schizophrenia especially when combined with psychosocial interventions that focus on function such as CBSST. Thus, we also propose to assess the tolerability and impact of CRT on patients with late-life schizophrenia.

DETAILED DESCRIPTION:
Eighty subjects will be randomized into 2 arms, CBSST Group and Treatment as Usual Group. Both Arms will run for a total of 52 weeks. The CBSST Group will attend 2-hour weekly sessions for 9 months and attend follow up assessments every 4 months. The Treatment as Usual Group will continue with their normal psychiatric treatment as usual and also attend follow up assessments every 4 months. After subjects in the Treatment as Usual Arm finish, they will continue on to the CBSST Group arm.

After the completion of the CBSST Group Arm, 24 subjects who are willing to consent to CRT will continue with an additional 2-hour weekly session of Cognitive Remediation Treatment for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and above.
* All races and ethnicities.
* Females and males.
* Meets DSM-IV TR criteria for a current diagnosis of schizophrenia, schizoaffective disorder, schizophreniform, delusional disorder, or psychotic disorder NOS.
* Clinically stable as operationalized by (1) having not been admitted to a psychiatric hospital within the 3 months prior to assessment, (2) having had no change in antipsychotic medication dosage within the 4 weeks prior to assessment, and (3) and ascertained to be clinically stable by one the study psychiatrists.
* Willingness and ability to speak English
* Willingness to provide informed consent
* Corrected visual ability that enables reading of newspaper headlines and corrected hearing capacity that is adequate to respond to a raised conversational voice.

Exclusion Criteria:

* Meets criteria for a cognitive disorder secondary to a neurological or other medical disorder affecting the ability to participate in CBSST.
* Diagnosis of bipolar disorder or current major depressive episode.
* Meets diagnostic criteria for substance use or dependence within the 6 months prior to the initial assessment except for caffeine or nicotine.
* Electroconvulsive Therapy (ECT) within 6 months of initial assessment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of CBSST in improving social function | At termination

CONTACTS AND LOCATIONS:
Overall Officials: David C. Mamo, MD, MSc, Principal Investigator — Centre for Addiction and Mental Health; Tarek Rajji, MD, FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rajji TK, Mamo DC, Holden J, Granholm E, Mulsant BH. Cognitive-Behavioral Social Skills Training for patients with late-life schizophrenia and the moderating effect of executive dysfunction. Schizophr Res. 2022 Jan;239:160-167. doi: 10.1016/j.schres.2021.11.051. Epub 2021 Dec 9. PMID 34896870
- [Derived] Gerretsen P, Voineskos AN, Graff-Guerrero A, Menon M, Pollock BG, Mamo DC, Mulsant BH, Rajji TK. Insight Into Illness and Cognition in Schizophrenia in Earlier and Later Life. J Clin Psychiatry. 2017 Apr;78(4):e390-e397. doi: 10.4088/JCP.16m10741. PMID 28297590
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital. It is fully affiliated with the University of Toronto, and is a PAHO/WHO Collaborating Centre. — http://www.camh.net/research